CLINICAL TRIAL: NCT01934257
Title: The Evaluation of Infant Formulas Fed to Infants With Common Feeding Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 3332-5
Record Dates: First submitted 2013-08-27; First posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Common Infant Feeding Problems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Marketed milk-based lactose-containing infant formula (Other)
  Interventions: Other: Marketed milk-based lactose-containing infant formula
- Marketed milk-based lactose-free infant formula (Other)
  Interventions: Other: Marketed milk-based lactose-free infant formula
- Marketed soy-based lactose-free infant formula (Other)
  Interventions: Other: Marketed soy-based lactose-free infant formula

INTERVENTIONS:
Other: Marketed milk-based lactose-containing infant formula
  Arms: Marketed milk-based lactose-containing infant formula
Other: Marketed milk-based lactose-free infant formula
  Arms: Marketed milk-based lactose-free infant formula
Other: Marketed soy-based lactose-free infant formula
  Arms: Marketed soy-based lactose-free infant formula

SUMMARY:
This clinical trial will determine if the formula given to infants experiencing fussiness, crying, cramping, gas, and/or diarrhea, is accepted and well tolerated and helps to resolve symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 2 and 12 weeks of age
* Subject has currently been receiving a milk-based lactose-containing formula for at least 5 days as the sole item of diet
* Subject has never switched to any lactose free formula
* The parent/guardian who will fill out the quality of life questionnaire is female and at least 18 years of age
* The parent/guardian has reported an unsolicited history of feeding problems including fussiness/crying/cramping, gas, or diarrhea
* Signed Informed Consent

Exclusion Criteria:

* Subject is in daycare for more than 4 hours per day (20 hours per week)
* Subject has serious perinatal complications, underlying disease or congenital malformations that impair normal formula feeding
* The parent/guardian who will fill out the quality of life questionnaire has chronic illness, e.g. diabetes, inflammatory bowel disease or other illness requiring daily medication or treatment
* Subject has acute infectious diarrhea or any other intercurrent illness

Ages: 2 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 296 (Actual)
Dates: Start 1994-06; Primary Completion 1996-06 (Actual); Study Completion 1996-06 (Actual)

PRIMARY OUTCOMES:
Early Infant Temperament Questionnaire | 14 days

SECONDARY OUTCOMES:
Infant Characteristic Questionnaire | 14 days
Maternal Efficacy Questionnaire | 14 days
Mental Health Inventory Questionnaire | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Colin Rudolph, M.D., Ph.D, Study Director — Mead Johnson & Company
Locations (19):
- United States (18):
  - Dr. Mark Pearlman, Aurora, California
  - Gould Medical Foundation, Modesto, California
  - Memorial Medial Center Research, Savannah, Georgia
  - Welborn Clinic Peds, Evansville, Indiana
  - Riveria Pediatrics, Indianapolis, Indiana
  - Kentucky Pediatrics, Bardstown, Kentucky
  - Kids Med South, Baton Rouge, Louisiana
  - The Pediatric Group, Princeton, New Jersey
  - Chapel Hill Pediatrics, Durham, North Carolina
  - Henderson Pediatrics, Fletcher, North Carolina
  - Matthews Children Group, Matthews, North Carolina
  - Capital Pediatrics, Raleigh, North Carolina
  - Pediatric Medical Associates, Havertown, Pennsylvania
  - Pennridge Pediatrics, Sellersville, Pennsylvania
  - Pittsburgh Pediatric Research, Upper Saint Clair, Pennsylvania
  - Lewis Gale Clinic, Salem, Virginia
  - Vancouver Clinic, Vancouver, Washington
  - Rhinelander Medical Center, Rhinelander, Wisconsin
- Dr. David Conner, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Sherman AL, Anderson J, Rudolph CD, Walker LS. Lactose-Free Milk or Soy-Based Formulas Do Not Improve Caregivers' Distress or Perceptions of Difficult Infant Behavior. J Pediatr Gastroenterol Nutr. 2015 Jul;61(1):119-24. doi: 10.1097/MPG.0000000000000743. PMID 25643020